CLINICAL TRIAL: NCT00876928
Title: Effect of Vitamin D Supplementation on Pre-Diabetes in a Minority Population
Brief Title: Vitamin D in Minorities With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Mayer Davidson, Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Vitamin D-Prediabetes; 1-09-CR-15 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-04

CONDITIONS: Pre-diabetes
Keywords: pre-diabetes; minorities; oral glucose tolerance test; disposition index; insulin secretion; insulin sensitivity; diabetes
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Diabetes Mellitus | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects with low vitamin D levels and pre-diabetes
  Interventions: Drug: placebo
- vitamin D (Experimental): Subjects with low vitamin D levels and pre-diabetes
  Interventions: Drug: vitamin D

INTERVENTIONS:
Drug: vitamin D — liquid vitamin D3 dissolved in medium chain triglyceride once a week
  Arms: vitamin D
Drug: placebo — medium chain triglyceride given once per week
  Arms: Placebo

SUMMARY:
Vitamin D supplementation in minority subjects with both pre-diabetes and low vitamin D levels will delay the development of diabetes.

DETAILED DESCRIPTION:
Low vitamin D levels 1) are associated with abnormalities in insulin secretion and insulin action, 2) predict the development of diabetes in those without diabetes, and 3) are more common in people with diabetes. Minority populations (African-Americans and Latinos) are more likely to have both low levels of vitamin D and diabetes. This study will identify minority individuals who are at increased risk for diabetes (those with central obesity, family history of diabetes in first degree relatives and either with hypertension or being treated for hypertension), and determine if they have both pre-diabetes, ie, impaired fasting glucose and/or impaired glucose tolerance, and low levels of vitamin D. Those that have both will be randomized to either high doses of vitamin D or placebo and insulin secretion and action as well as changes in the oral glucose tolerance test (reversion to normal, maintenance of pre-diabetes or development of diabetes) will be monitored at 3 month intervals for one year. This study will test the hypothesis that the increased amount of diabetes in minority populations may be due in part to low levels of vitamin D and whether supplementing this vitamin may delay the development of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 40.
2. Impaired fasting glucose (FPG level greater than 100 and less than 126 mg/dl); and/or
3. Impaired glucose tolerance (2-h plasma glucose concentration after 75 gram glucose load greater than 140 and less than 200 mg/dl)
4. Serum 25-OHD less than 30 ng/ml
5. Able and willing to provide informed consent

Exclusion Criteria:

1. FPG greater than 126 mg/dl or 2-hour-OGTT plasma glucose greater than 200 mg/dl
2. Major psychiatric disorder on medication (excluding successfully treated depression)
3. Diagnosed diabetes mellitus
4. HIV/AIDS
5. Major hematological, hepatic (AST/ALT levels greater than or equal to 2 times normal) or renal eGFR less than 60 ml/min) disorder
6. History of carcinoma, except skin basal cell or squamous cell skin carcinomas
7. Heart failure, unstable angina or history of a myocardial infarction
8. Alcohol or substance abuse
9. Current treatment with glucocorticoids
10. Current treatment with diabetes medications, including metformin
11. Cushing's syndrome
12. Primary hyperparathyroidism
13. Nephrolithiasis
14. Pregnancy or breast-feeding
15. Regular visits to a tanning salon (unlikely in this minority population)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayer B. Davidson, MD, Principal Investigator — Charles Drew University
Locations (1):
- Charles Drew University, Los Angeles, California, United States

REFERENCES:
- [Derived] Sinha-Hikim I, Duran P, Shen R, Lee M, Friedman TC, Davidson MB. Effect of long term vitamin D supplementation on biomarkers of inflammation in Latino and African-American subjects with pre-diabetes and hypovitaminosis D. Horm Metab Res. 2015 Apr;47(4):280-3. doi: 10.1055/s-0034-1383652. Epub 2014 Jul 10. PMID 25011019
- [Derived] Davidson MB, Duran P, Lee ML, Friedman TC. High-dose vitamin D supplementation in people with prediabetes and hypovitaminosis D. Diabetes Care. 2013 Feb;36(2):260-6. doi: 10.2337/dc12-1204. Epub 2012 Oct 1. PMID 23033239

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: Subjects with low vitamin D levels and pre-diabetes
  Liquid vitamin D3 dissolved in medium chain triglyceride once per week
Period: Overall Study
Arm/Group | Placebo | Vitamin D
Started | 56 | 61
Completed | 53 | 56
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 2 | 5
Not completed — Hypokalemia-affects insulin secretion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Total
Number analyzed (Participants) | 56 | 61 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 55 | 107
  >=65 years | 4 | 6 | 10
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (7.0) | 52.3 (8.0) | 52.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 79
  Male | 20 | 18 | 38
Region of Enrollment [Number; unit: participants]
  United States | 56 | 61 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Develop Diabetes
Description: Diabetes defined by a FPG>=126 mg/dl or a 2-hr glucose concentration on an OGTT of >=200 mg/dl
Time Frame: one year
Population: Minorities with pre-diabetes and hypovitaminosis D
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 53 | 56
percentage of participants | 9 | 12
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; Null hypothesis is that there is no effect of vitamin D on the development of diabetes in people with pre-diabetes and hypovitaminosis D. There were no published data when this trial was started on the effect of vitamin D in pre-diabetes making a power calculation difficult; Test type: Superiority or Other; p = 0.61, Chi-squared — A chi square test was used for the number of participants developing diabetes and a 2-way repeated measures ANOVA for the disposition index; Percent of patients developing diabetes = 10, 95% CI 2-sided [8 to 12] — Primary outcome compared the number of participants developing diabetes after receiving vitamin D or placebo for one year. Secondary outcome compared changes in 2-way repeated measures ANOVA; therefore,no confidence intervals/dispersion parameters

2. Secondary Outcome: Disposition Index
Description: Measure of insulin secretion multiplied by measure of insulin sensitivity,both derived from oral glucose tolerance test; higher values are better
Time Frame: Baseline, 3, 6, 9, 12 months
Population: modified intent to treat
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 53 | 56
Unitless
  Dispostion Index at baseline | 1.4 (0.5) [1.3 to 1.6] | 1.3 (0.4) [1.2 to 1.3]
  Disposition Index at 3 months | 1.5 (0.8) | 1.3 (0.5)
  Disposition Index at 6 months | 1.4 (0.6) | 1.2 (0.5)
  Disposition Index at 9 months | 1.3 (0.6) | 1.3 (0.4)
  Disposition Index at 12 months | 1.6 (1.6) | 1.3 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D; The null hypothesis is that there would be no difference in the changes in the Disposition Index between the 2 groups over the year; Test type: Superiority or Other; p = 0.39, ANOVA

ADVERSE EVENTS:
Arm/Group | Placebo | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/56
Other Adverse Events (participants affected / at risk) | 0/53 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No